CLINICAL TRIAL: NCT02649101
Title: Thalidomide Plus Chemotherapy Versus Chemotherapy Alone: A Phase II Study in Advanced Breast Cancer
Brief Title: Thalidomide Plus Chemotherapy Versus Chemotherapy Alone for Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, LeiLei, Dr., Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZCHBC-007
Record Dates: First submitted 2015-12-13; First posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- thalidomide plus chemotherapy (Experimental): thalidomide tablet 100mg qn po
  Interventions: Drug: Thalidomide; Drug: Physician's choice chemotherapy
- chemotherapy (Active Comparator): Physician's choice chemotherapy. No constraints of the choice of chemotherapy drugs and regimens.
  Interventions: Drug: Physician's choice chemotherapy

INTERVENTIONS:
Drug: Thalidomide — Thalidomide tablet 100mg qn po.
  Other Names: Contergan
  Arms: thalidomide plus chemotherapy
Drug: Physician's choice chemotherapy — Investigators will declare no constraint of regimens.
  Other Names: no other name

SUMMARY:
Sixty advanced breast cancer patients are planed to enrolled in this clinical trial. Forty patients are enrolled into thalidomide plus chemotherapy group. Twenty patients are enrolled into chemotherapy alone group. There is no restriction on chemotherapy regimen and lines.

DETAILED DESCRIPTION:
The study compares the combination of thalidomide and chemotherapy with chemotherapy alone for the treatment of stage IV breast cancer. Efficacy and safety of the chemotherapy-thalidomide combination will be evaluated. Assessing the isolated effects of thalidomide in a setting where pre and post treatment serum specimens can be obtained will provide essential information about the mechanisms by which vascular endothelial growth factor(VEGF) inhibition affects tumor growth, and represents an ideal opportunity to evaluate the molecular effects of thalidomide on breast tumor.

ELIGIBILITY:
1. inclusion criteria:

   * Women >/= 18 and < 65 years of age .
   * Histologically or cytologically confirmed breast cancer with evidence of metastatic disease. (Note: the participant must be recovered from any clinically significant toxicity thereof last therapy.)
   * ECOG performance status 0-2.
   * Adequate bone marrow, kidney and liver function.
   * ER/PR breast cancer positive patients must have received and progressed on at least one endocrine therapy (adjuvant or metastatic), or have disease that the treating physician believes to be inappropriate for endocrine therapy.
2. exclusion criteria:

   * Prior treatment with thalidomide.
   * Patients with HER2 positive disease.
   * Untreated and/or uncontrolled brain metastases.
   * Prior malignancy unless curatively treated and disease-free for > 5 years prior to study entry. Prior adequately treated non-melanoma skin cancer, in situ cancer of the cervix, DCIS or stage I grade 1 endometrial cancer allowed.
   * Known HIV (Human Immunodeficiency Virus) infection.
   * Pregnant or breast-feeding women.
   * Bilateral invasive breast cancer.
   * Cardiac and thrombotic disease or risk for same as judged by Investigator.
   * Other serious illness or medical conditions such as (partial list- review with Investigator) history of significant neurologic or psychiatric disorders that would prohibit the understanding and giving of informed consent, active uncontrolled infection, active peptic ulcer, unstable diabetes mellitus or subjects with symptomatic, intrinsic lung disease resulting in dyspnea at rest.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) | Change from Baseline RECIST at 6 months was assessed every 6 weeks up to 24 weeks. Data collection is from date of randomization until the date of first documented progression assessed up to 6 months.
  PFS is defined as the months that from the anticipation of the clinical-trial to the progress of breast cancer.

SECONDARY OUTCOMES:
Overall survival(OS) | Survival assessed every 8 weeks up to 100 months following objective disease progression. Data collection is from date of randomization until the date of death from any cause, assessed up to 100 months.
  OS is defined as the months that from the anticipation of the clinical-trial to the death of patients.

CONTACTS AND LOCATIONS:
Overall Officials: xiaojia wang, doctor, Study Chair — Director
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided